CLINICAL TRIAL: NCT03790020
Title: COMPARISON OF TRANSVERSUS ABDOMINIS PLANE BLOCK, LOCAL ANESTHETIC INJECTION TO THE PORT SITES AND INTRAPERITONEAL LOCAL ANESTHESIA APPLICATIONS IN POSTOPERATIVE PAIN MANAGEMENT IN PATIENTS WITH LAPAROSCOPIC APPENDECTOMY
Acronym: APPENDECTOMY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ANIL ERGIN.....
Record Dates: First submitted 2018-12-15; First posted 2018-12-31 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
Keywords: acute appendicitis; postoperative pain relief; local anesthetic; laparoscopic appendectomy
MeSH Terms: conditions — Pain, Postoperative; Appendicitis | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: 3 types of local anesthetic applying method will be compared
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- transversus abdominis plane Block (Active Comparator): Transversus abdominis plane block (10 cc / 10 cc, 0.5% bupivacaine to the right and left transversus abdominis muscle regions) will be applied.
  Interventions: Drug: Bupivacaine
- TROCHAR SITES LOCAL ANESTHETIC INJECTION (Active Comparator): local anesthetic injection (6 cc to subxiphoid and infraumbilical trocar sites, 4 cc instead of 2 cc, 0.5% bupivacaine solution to be applied)
  Interventions: Drug: Bupivacaine
- INTRAPERİTONEAL LOCAL ANESTHETIC SPREADING METHOD (Active Comparator): Intraperitoneal direct vision of the appendix excision area-periappendiciall area under the direct injection of local anesthetic spraying process (percutaneous method injected into the periappendicial area 1: 1 diluted with 20 cc SF, 20 cc 0.5% bupivacaine solution total 40 cc spraying will be applied.
  Interventions: Drug: Bupivacaine
- CONTROL GROUP (No Intervention): group will be the control group and any of these methods will not be applied,

INTERVENTIONS:
Drug: Bupivacaine — In our study this local anesthetic agent will be applied for postoperative pain relief
  Other Names: marcaine
  Arms: INTRAPERİTONEAL LOCAL ANESTHETIC SPREADING METHOD; TROCHAR SITES LOCAL ANESTHETIC INJECTION; transversus abdominis plane Block

SUMMARY:
The most important determinant of the recovery in abdominal surgery is postoperative pain. Postoperative pain can be explained by 2 pathways connected to the peritoneum; The first is the parietal peritoneum, whose innervation is very rich and the other is the visceral peritoneum which is stimulated at the vagus level. Since 1950, they have been injecting local anesthetic for post-surgery pain. inflammation and peritoneal irritation are the most important factors of pain when acute appendicitis is diagnosed. . This increases the length of hospital stay and increases the cost of pain relief, and reduces patient satisfaction. The aim of this study is to evaluate the application of Transversus Abdominis Plane Block . local anesthetic injection to the port sites, intraperitoneal periappendiceal local anesthetic injection is compared with the control group without any local anesthetic application to investigate which group has more analgesic effectiveness and thus reduce the amount of analgesics needed postoperatively, hospitalization Shortening the duration of the patient and taking the patient comfort to the next level.

DETAILED DESCRIPTION:
Laparoscopic Appendectomy procedure will be performed in patients over 18 years of age who are hospitalized from the emergency department for acute appendicitis. 4 patient group will be established. The number of samples determined for Power: 0.80 and alpha: 0.05 was determined as minimum n: 28 for each group. Therefore, the groups will be determined to include 28 patients. In our clinic, local anesthetic injection to the trocar areas is routinely performed in laparoscopic appendectomy operations. After endotracheal intubation at the beginning of the operation, after appropriate skin staining and sterile dressing Transversus abdominis plane block (10 cc / 10 cc, 0.5% bupivacaine to the right and left transversus abdominis muscle regions) will be applied. local anesthetic injection to the pre-incision trocar sites (8 cc instead of infraumbilical trocar, 6 cc instead of the other 2 trocar 20 cc 0.5% bupivacaine solution will be applied), following intraperitoneal direct visualization of the appendiceal region - local anesthetic spraying into the periappendiceal area(1: 1 diluted with 20 cc saline, 20 cc 0.5% bupivacaine solution total 40 cc spraying ) will be applied. The fourth group will be the control group and any of these methods will not be applied, operation time and peroperative complications (appendiceal perforation etc.) will be recorded.Paracetamol 1 g + 1 mg / kg tramadol IV will be applied to all four groups as standard before extubation. Visual analogue scale (VAS) will be applied to all patients in the postoperative period. If VAS> 3 is still present, a dose of 1 mg / kg tramadol will be administered. Tenoxicam 1x1 IV will be applied to the patients on the 12th hour. All patients were postoperative; 1,2,4,6,12,24. VAS scores , patient satisfaction (0: never satisfied, 5: very satisfied) will be recorded. The group of patients will be determined according to the order of surgery. Pain scores of the patients will be performed by a physician who is not in the operation who does not know which group is taken. The patients included in the group will not be known to the patient by the pain scoring system and the study will be done as double blind. Patients will be randomized with this method.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with acute appendicitis in emergency department

Exclusion Criteria:

* Patients who have to undergo peroperative open appendectomy procedure.
* Patients with local anesthetic or non steroid antiinflammatory allergy
* Patients in pregnancy
* Patients with connective tissue disease
* Patients with malignancy detected in pathological examination of postoperative appendix and patients with any malignancy diagnosis
* Perforated patients peroperatively
* Patients who were evaluated as plastron appendicitis peroperatively

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
compare of local anesthetic applying methods for postoperative pain relief by VAS (Visual Analog Scala) | 24 hours
  pain scores of the participants will be followed at postoperative 1,2,4,6,12,24 hour (up to 24 hours).
  (VAS: from 0 to 10, 0 = no pain, 10 = the worst pain) The higher score idicates the worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No